CLINICAL TRIAL: NCT05103072
Title: Subthalamic Nucleus Stimulation With Directional Leads on Patients With Parkinson Disease at Fluctuations and Dyskinesia Stage
Acronym: NSTBOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2021_843_0162
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Parkinson Disease; Subthalamic Nucleus Stimulation; Directional Electrodes
Keywords: Parkinson Disease; Subthalamic nucleus stimulation; directional electrodes
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- testing all the plots: the investigator chose the best plot of the leads for stimulation by a procedure long and exhausting for the patient and the examinator (" plot by plot ")
- Guide X Software: the investigator can chose the plot using a software (Guide Xt), which can delete the exhausting test

SUMMARY:
Patients with subthalamic nucleus have to go through a lot of examinations and tests, before and after surgery which is difficult, sometimes painful, for the patient.

The investigators used to chose the best plot of the leads for stimulation by a procedure long and exhausting for the patient and the examinator.

The investigators can chose the plot using a software (Guide Xt), which can delete the exhausting test.

The investigators would like to study the non inferiority of this tool to choose the best plot .

ELIGIBILITY:
Inclusion Criteria:

* age : >18Y
* All patient with Parkinson disease eligible for sub thalamic surgery (CAPSIT criterias) in CHU AMIENS

Exclusion Criteria:

* patient doesn't consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is a non interventional retrospective study. Data were collected before and after surgery of subthalamic nucleus stimulation of patients with Parkinson Disease.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Estimated)
Dates: Start 2021-09-21 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Increase of MDS UPDRS 3 score | 3 months
  The MDS-UPDRS was developed to evaluate various aspects of Parkinson's disease including non-motor and motor experiences of daily living and motor complications.
  The MDS-UPDRS has four parts, namely, I: Non-motor Experiences of Daily Living; II: Motor Experiences of DailyLiving; III: Motor Examination; IV: Motor Complications.Twenty questions are completed by the patient/caregiver. Item-specific instructions and an appendix of complementary additional scales are provided.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aubignat M, Berro A, Tir M, Lefranc M. Imaging-Guided Subthalamic Nucleus Deep Brain Stimulation Programming for Parkinson Disease: A Real-Life Pilot Study. Neurol Clin Pract. 2024 Dec;14(6):e200326. doi: 10.1212/CPJ.0000000000200326. Epub 2024 Sep 11. PMID 39282508